CLINICAL TRIAL: NCT05448846
Title: Effect of a Personalized Physical Exercise Program on Functional Capacity and Quality of Life in Older Colorectal Cancer Patients
Brief Title: Exercise Program for Colorectal Older Patients
Acronym: ECOOL
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital General Universitario Gregorio Marañon (Other)
Collaborators: Instituto de Salud Carlos III (Other Government)
Responsible Party: Principal Investigator, Dr. Jose Antonio SERRA-REXACH, Head Of Geriatry Department, Hospital General Universitario Gregorio Marañon
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: PI21/01729
Record Dates: First submitted 2022-06-10; First posted 2022-07-07 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Colorectal Neoplasms; Aged
Keywords: Cancer; Elderly; Exercise; Prehabilitation; Rehabilitation; Surgery; Colorectal; Physical activity
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasms; Motor Activity | interventions — Enhanced Recovery After Surgery

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator): Usual care (i.e., 'Enhanced Recovery After Surgery' (ERAS) protocol)
  Interventions: Procedure: Enhanced Recovery After Surgery
- Home-based multicomponent exercise program (Experimental): Complete a home-based multicomponent exercise program from diagnosis to 3 months after surgery in addition to ERAS protocol.
  Interventions: Procedure: Enhanced Recovery After Surgery; Behavioral: Home-based multicomponent exercise program (EXE)

INTERVENTIONS:
Procedure: Enhanced Recovery After Surgery — ERAS protocol includes preoperative counselling, optimization of nutrition, standardized analgesic and anesthetic regimens and early mobilization.
  Other Names: ERAS
Behavioral: Home-based multicomponent exercise program (EXE) — Home-based multicomponent exercise program:
  A) Strength and balance (20 to 40 minutes, 2 days/week):
  * Chair sit to stand exercise | 1 to 3 sets completing repetitions until rating 5 to 8 in the Rated of Perceived Exertion, 0-10 scale (RPE).
  * Seated curl to press exercise | 1 to 3 sets completing repetitions until rating 5 to 8 RPE.
  * Monopodal balance | 1 to 3 sets with progressive time targets up to 60-second for each leg.
  B) Gait (at least 30 minutes at an intensity that allows for comfortable conversation, 2 days/week on separate days from strength and balance exercise)
  C) Inspiratory Muscle Training: 30 inspirations at 40% of maximal inspiratory pressure through a Power Breathe device, 2 times per day)
  Other Names: EXE
  Arms: Home-based multicomponent exercise program

SUMMARY:
The Exercise for COlorectal OLder patients (ECOOL program) is randomized controlled trial to assess the effects of an exercise program on physical function and health-related quality of life of patients 75 years and older with colorectal cancer undergoing surgery. ECOOL is a multicomponent home-based exercise intervention focused on the development of strength, balance, gait ability and inspiratory muscle function of older patients who receive weekly telephone follow-up from cancer diagnosis to 3 months after surgery. The investigators expect that ECOOL program will improve physical function and health-related quality of life of older patients 3 months after surgery and to maintain these benefits up to 6 months after surgery compared with the control group receiving usual care.

DETAILED DESCRIPTION:
Colorectal cancer (CRC) is the second most common cancer and the second cause of cancer-related death in Europe. Thirty-one percent of new cases are older than 74 years. The decrease in reserve capacity (i.e., frailty), comorbidity and the surgical treatment imply that the elderly patient is at greater risk of functional decline (reported between 15% and 18% three months after surgery).Up to 50% of those who have experienced functional decline do not recover previous levels of functional independence. The aim of this research is to investigate the effects of a multicomponent physical exercise program on physical function and health-related quality of life (HRQoL) of patients 75 years and older with CRC undergoing surgery. The exercise program focuses on the development of strength, balance, gait ability and inspiratory muscle function of older patients who receive weekly telephone follow-up from cancer diagnosis to 3 months after surgery. Weekly telephone follow-up is provided by an exercise specialist who monitors adherence to the exercise program and insists on its compliance, clarifies any doubt and prescribes exercise progression. Moreover, patients complete a supervised exercise session at baseline, during hospitalization and one month after surgery to ensure correct exercise execution and provide feedback. The investigators expect that ECOOL program will improve physical function and HRQoL of older patients 3 months after surgery and to maintain these benefits up to 6 months after surgery compared with the control group receiving usual care.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 75 years or older diagnosed with colorectal cancer.
* Patients included in colorectal surgery waiting list of the Hospital General Universitario Gregorio Marañon (Madrid, Spain)
* Patients able to communicate, understand and sign the informed consent.

Exclusion Criteria:

* Patients finally excluded for colorectal surgery.
* Patients with absolute contraindications to exercise
* Walk disability (FAC <2)
* Severe cognitive impairment (MMSE <18)
* Terminal illness

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 252 (Estimated)
Dates: Start 2022-04-08 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in Health-related Quality of Life (HRQoL) of cancer patients | From baseline to 1 week, 3 months and 6 months after surgery
  HRQOL measured by the European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30). This questionnaire provides 0-100 scores in different single- or multi-item scales of three different domains of HRQoL:
  * Global health status (higher scores mean better health status)
  * Function (higher scores mean better function)
  * Symptomatology (higher scores mean worse symptomatology)
Change in supplementary HRQoL scales for colorectal cancer patients | From baseline to 1 week, 3 months and 6 months after surgery
  The European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire for Colorectal Cancer 29 (EORTC QLQ-CR29) will be employed. This questionnaire consists of 4 multi-item scales and 19 single-items assessing a range of symptoms and problems common among patients with colorectal cancer. All of the scales and single-item measures range in score from 0 to 100. A high score for the functional scale and functional single-items represents a high level of functioning, whereas a high score for the symptom scales and symptom single-items represents a high level of symptomatology or problems.
Change in supplementary HRQOL scales for elderly cancer patients | From baseline to 1 week, 3 months and 6 months after surgery
  The European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire for Elderly cancer patients (EORTC QLQ-ELD14) will be employed. The EORTC QLQ-ELD14 contains important age-specific issues for elderly cancer patients, which was developed to supplement the EORTC QLQ-C30. The QLQ-ELD14 comprises 14 items, made up of 5 scales (mobility, worries about others, future worries, maintaining purpose and burden of illness) and 2 single items (joint stiffness and family support). Scores in all areas range from 0 to 100, with higher scores indicating worse QoL in the case of mobility, joint stiffness, worries about others, future worries, and burden of illness, and better QoL in family support (feel able to talk to the family about the illness) and maintaining purpose.
Change in functional capacity | From baseline to 1 week, 3 months and 6 months after surgery
  Change in functional status measured by Barthel Index. This index measures the extent to which somebody can function independently and has mobility in their activities of daily living (ADL). Including: feeding, bathing, grooming, dressing, bowel control, bladder control, toileting, chair transfer, ambulation and stair climbing. Scoring 0 points would be dependent in all assessed activities of daily living, whereas a score of 100 would reflect independence in these activities. Low scores on individual items highlight areas of need.

SECONDARY OUTCOMES:
Change in physical function | From baseline to admission for surgery and at 1, 3 and 6 months after surgery
  Changes in physical function measured by the Short Physical Performance Battery (SPPB). SPPB consists of 3 components: standing balance, gait speed, and repeated chair rise. Balance includes standing with feet side-by-side, semi-tandem, and tandem stance. Gait speed scores reflected the time needed to walk 4 m. Repeated chair rise is scored based on time to complete 5 chair rises. Each SPPB component is scored from 0 to 4, and the total sore ranged was 0-12 with higher scores indicating better function.
Change in frailty status | From baseline to admission for surgery and at 1, 3 and 6 months after surgery
  Changes in frailty status measured by the Fried's phenotype. This method classifies older adults as frail, pre-frail or non-frail based on five criteria: I) Weight loss (unintentionally), II) Exhaustion, III) Low physical activity, IV) Low habitual gait speed and V) Low handgrip strength.
Change in upper limb muscle size (thickness, mm) | From baseline to admission for surgery and at 1, 3 and 6 months after surgery
  Ultrasound-based determination of biceps brachialis muscle thickness
Change in lower limb muscle size (thickness, mm) | From baseline to admission for surgery and at 1, 3 and 6 months after surgery
  Ultrasound-based determination of rectus femoris muscle thickness
Change in inspiratory muscle function | From baseline to admission for surgery and at 1, 3 and 6 months after surgery
  Measurement of the maximum static inspiratory pressure (cm H2O) that a subject can generate at the mouth (PImax). This measure reflects the inspiratory muscle function (strength)
Change in physical fitness | From baseline to admission for surgery and at 1, 3 and 6 months after surgery
  Change in physical fitness evaluated through a modified version of the Senior Fitness Test (Rikli & Jones, 2001) designed to assess different components of older adults physical fitness:
  * Upper and lower limbs muscle strength (30 seconds arm curl test and 30 second Sit to Stand tests, in number of repetitions)
  * Upper and lower limbs flexibility (Back Scratch test and Chair Sit and Reach test, centimeters)
  * Monopodal Static Balance (Flamingo test, in seconds)
  * Agility (8-foot Timed Up&Go test, in seconds)
  * Maximal gait speed (30-meter maximal walking speed test, in meters per second)
  * Cardiorespiratory fitness (2-minute step test, in number of steps)
  The raw values obtained in each test will be expressed in specific normative values (percentiles) for the non-institutionalized Spanish elderly (Pedrero-Chamizo, 2012). Finally, a single measure of physical fitness will be reported by averaging the percentile values obtained for all test.
Change in physical activity | From baseline to admission for surgery and at 1, 3 and 6 months after surgery
  Change in physical activity evaluated through the Physical Activity Scale for Elderly (PASE).This questionnaire is comprised of self-reported occupational, household and leisure activities items over a one-week period that provides a global score ranged from 0 (no physical activity) to 400 or more (more physical activity)
Comprehensive Complication Index (CCI) | within a 90 days postoperative time period
  The Comprehensive Complication Index (CCI) is calculated as the sum of all Clavien-Dindo complications that are weighted for their severity. The final formula yields a continuous scale that ranks the cumulative burden from any combination of complications from 0 (no complication) to 100 (death) with higher values indicating a higher cumulative burden in a single patient.
Length of stay in hospital after colorectal surgery (days) | From hospital admission for colorectal surgery up to discharge after surgery assessed up to 12 months.
  Duration in days
Prevalence of Anxiety and Depression | At baseline and at 1, 3 and 6 months after surgery
  Assessed by the Hospital Anxiety and Depression Scale (HADS). This scale consisted of 14 items that evaluate anxiety (7 items, 28 points) and depression (7 items, 28 points).For each mood disorder, scores greater than 10 are considered indicative of morbidity. A score of 8-10 is interpreted as borderline, and scores below 8 indicate no significant morbidity.
Prevalence of cancer-cachexia | At baseline and at 1, 3 and 6 months after surgery
  Prevalence of cancer-cachexia measured by the definition and classification of cancer cachexia: An international consensus (Fearon et al. 2012)
Prevalence of sarcopenia | At baseline and at 1, 3 and 6 months after surgery
  Prevalence of sarcopenia defined by the 'European Working Group on Sarcopenia in Older People 2' criteria
Number of hospital readmissions | From baseline to 3 and 6 months after surgery
  Number and mean length of hospital readmissions during the follow-up
Rate of mortality | From baseline to 6 month after surgery
  All-cause mortality

OTHER OUTCOMES:
Number of pre-operative comorbidities | Baseline
  Charlson Comorbidity Index
Pre-operative physical status classification | Baseline
  American Society of Anesthesiologists (ASA) physical status classification system. This scale consists of 6 different levels, from I (normal healthy patient) to VI (a declared brain-dead patient whose organs are being removed for donor purposes)
Number of pre-operative geriatric syndromes | Baseline
Type of adjuvant treatment | From baseline to 6 months after colorectal surgery
  Type of adjuvant treatment(s) received (ie., radiotherapy, chemotherapy or immunotherapy)
Dose of adjuvant treatment | From baseline to 6 months after colorectal surgery
  Total dose of adjuvant treatment(s) received
Colorectal Surgery Procedure | Immediately after the colorectal surgery
  Type of colorectal surgery procedure (i.e., open surgery or laparoscopic)

CONTACTS AND LOCATIONS:
Overall Officials: Jose Antonio Serra-Rexach, PhD, MD, Principal Investigator — HGU Gregorio Marañon
Locations (1):
- Hospital general Universitario Gregorio Marañón, Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial will be shared after deidentification. The disclosure of individual patient data must be in compliance with the provisions of the Organic Law on Data Protection and Digital Rights of the Government of Spain (Ley Orgánica 3/2018, de 5 de diciembre, de Protección de Datos Personales y garantía de los derechos digitales).
Supporting Information: Study Protocol, ICF
Time Frame: Data will be available from 3 months to 5 years following article publication.
Access Criteria: Data will be shared only to Investigators whose proposed use of the data has been approved by an independent review committee ("learned intermediary") identified for this purpose. Proposals should be directed to joseantonio.serra@salud.madrid.org. To gain access, data requestors will need to sign a data access agreement.

REFERENCES:
- [Derived] Macias-Valle A, Rodriguez-Lopez C, Gonzalez-Senac NM, Mayordomo-Cava J, Vidan MT, Cruz-Arnes ML, Jimenez-Gomez LM, Dujovne-Lindenbaum P, Perez-Menendez ME, Ortiz-Alonso J, Valenzuela PL, Rodriguez-Romo G, Serra-Rexach JA. Exercise effects on functional capacity and quality of life in older patients with colorectal cancer: study protocol for the ECOOL randomized controlled trial. BMC Geriatr. 2023 May 22;23(1):314. doi: 10.1186/s12877-023-04026-6. PMID 37211611